CLINICAL TRIAL: NCT04001296
Title: A Study to Examine the Impact of a 21day School Brushing Intervention on the Knowledge, Behaviour and Oral Health of School Children
Brief Title: The Impact of a 21day School Brushing Intervention on the Knowledge, Behaviour and Oral Health of School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: World Dental Federation (FDI) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FDIUL-BDN-2018-01
Record Dates: First submitted 2019-06-25; First posted 2019-06-28 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Dental Plaque; Behavior; Behavior, Health
Keywords: Behavior; Toothbrushing; Toothpastes; Dental Caries; Education, Dental
MeSH Terms: conditions — Dental Plaque; Behavior; Health Behavior; Dental Caries

STUDY DESIGN:
Intervention Model Description: This study is a two-arm, parallel, stratified, cluster randomised trial. Clusters in this study are infant / junior schools in Indonesia and Nigeria. Ten schools in each country will be recruited. Schools will be matched into pairs by location (urban, semi-urban, rural) and then randomised to the 'intervention' and 'control' groups. using a randomisation table.
Who Masked: Outcomes Assessor
Masking Description: The data analysts / statisticians will not know whether the data they are analysing is from children in an Intervention or a Control school
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 21 day Brush Day and Night intervention (Experimental): The 21 day Brush Day and Night programme aims to instruct on and encourage twice a day brushing with a fluoridated toothpaste.
  Interventions: Behavioral: 21 day Brush Day and Night school programme
- Control schools (No Intervention): Schools / children who receive only toothpaste / toothbrushes, no 21 day Brush Day and Night intervention

INTERVENTIONS:
Behavioral: 21 day Brush Day and Night school programme — Children participating in the 21 day Brush Day and Night school programme are provided with toothpaste and a toothbrush each and enjoy brushing instruction, supervised brushing, and the singing of songs to facilitate learn the importance of brushing day and night, and stickers and calendars to track progress. A celebration is held at the end of the programme with certificates and rewards. The programme is supported by colourful and attractive materials with bespoke cartoon characters. Parents are provided with educational leaflets.
  Arms: 21 day Brush Day and Night intervention

SUMMARY:
In this study we aim to study the effectiveness of a specially designed 21 day Brush Day and Night programme for school children aged 6-9 which aims to establish the habit of twice a day toothbrushing for oral health.

The 21 day programme is led primarily by teachers with support from a oral health care professional.

Schools will be recruited in Indonesia and Nigeria to take part in the study. Half of the schools will run the 21 day programme with their children in school grades 1 to 3, half will act as a control.

DETAILED DESCRIPTION:
Background The World Health Organization reports that dental cavities affect 60-90% of children globally. FDI World Dental Federation and Unilever Oral Care have developed public health programmes to improve brushing habits over their 12-year partnership. The last of these (Phase III) named Brush Day & Night aimed to educate children in brushing twice daily with a fluoride toothpaste and gave useful information for a new project, Phase IV. The 21-day Brush Day & Night programme is an intense education activity designed to establish the habit of brushing day and night with a fluoride toothpaste. The programme involves daily brushing instruction and includes free toothpaste and toothbrushes.

Objective In Phase IV of the partnership, the aim is to evaluate the impact on the knowledge, behaviour and toothbrushing habits in schoolchildren aged 6-9 years old, after a 21-day school programme and compare with baseline and a control group. The enduring nature of the programme will be determined by the inclusion of 8 and 24-week time points.

Methods The study is a two-arm superiority randomized controlled trial. Clusters in this study are infant and junior schools in Indonesia and Nigeria. The study aims to recruit 20 schools, with children aged 6-9 years old, in each country.

At baseline, children in both intervention and control schools will answer a questionnaire and have their clinical oral health assessed using the Simplified Oral Hygiene Index (OHIs) and Decayed Missing and Filled Teeth (DMFT) index.

Children in the intervention schools will then take part in a structured 21-day Brush Day & Night intervention.

Children in the control schools will be provided with free toothpaste and toothbrushes but will not receive the 21-day intervention.

The questionnaires and OHIs assessment are repeated after the 21 days programme is completed and then again at 8 weeks and 24 weeks later for all participating children.

Parents/Carers/Guardians of all children will sign the informed consent and complete questionnaires on their own experience and attitudes to oral health and toothbrushing routine at each of the four times points (baseline, 21-day, 8 weeks and 24 weeks).

The study will be conducted by the National Dental Associations of Indonesia and Nigeria and was approved by the Ethics Committees of both countries.

Results:

The study is ongoing. Recruitment of schools started in Indonesia in February 2018 and in Nigeria in April 2018 for the first part of the study. This concluded in Indonesia in September 2018 and in Nigeria in November 2018. The second part of the study (the second half of the schools) started in November 2018 in Indonesia and December 2018 in Nigeria.

Conclusions:

The Investigators expect to collect all the data during 2019 and publish findings from the study by Q3 2020.

ELIGIBILITY:
Inclusion Criteria:

* Children aged in school year grades 1,2 and 3 years, aged 6-9 years
* Be of either gender and in good general health
* Be willing and be able (e.g. to brush teeth and understand and respond to questions) to participate in a 21-day Brush Day and Night activity at school and at home.
* Planning on attending their currently registered school for at least the next seven months.

Exclusion Criteria:

* Failure of the parent/carer/guardian to provide written informed consent.
* Subjects scheduled for medical or dental procedures during the duration of the study.
* Children who have a known allergy to any toothpaste ingredients
* Obvious signs of gross or untreated caries or of significant periodontal disease which in the opinion of the Dentist would affect the scientific validity of the study, or if the subject were to participate in the study would affect their wellbeing.
* Children or their family should have no affiliation (e.g. employee) with either the FDI or Unilever.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2020 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Change in reported brushing frequency and improved knowledge on recommendation to use fluoridated toothpaste | Baseline, 21 days, 8 weeks, 24 weeks
  Self-reported brushing frequency (no. of times a day) and time of day (morning / evening / other). Positive responses on use of a fluoridated toothpaste.

SECONDARY OUTCOMES:
Change in visible plaque and debris on teeth | Baseline, 21 days, 8 weeks, 24 weeks
  To measure the impact on oral health via plaque levels at baseline and after a 21-day school programme, 8 and 24 weeks later and compare with children and compare with children in the control group. Changes from Baseline will also be made Oral Health will be assessed by measuring plaque levels via the plaque levels via the Oral Hygiene Simplified Index (OHIs).

OTHER OUTCOMES:
Alterations in brushing frequency continue beyond the end of the 21 day programme. | 8 weeks and 24 weeks
  To evaluate the longer-term impact of the 21-day programme on knowledge/behaviour and oral health in children and knowledge/behaviour of their parents/carers after a period 8 weeks and 24 weeks (i.e. approx.. 7 months altogether). For the children, use of a questionnaire and plaque levels compared with baseline and after 21 days.
  For their parents/carers use of a questionnaire alone
The intervention influences the behaviour of parents / carers | Baseline, 21 days, 8 weeks, 24 weeks
  To provide evidence that the 21-day school program is effective in getting parents and carers to also improve their brushing habits and to brush day and night. Assessed via use of a questionnaire and compared with baseline and compared with parents/carers in their control group.
Children and adults who brush more frequently report a change in their own wellbeing | Baseline, 21 days, 8 weeks, 24 weeks
  Use of a simple 4 point scale with faces which signify different emotional states from happy to sad, compared with baseline and compared with children, parents/carers in their control group.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Melo, Prof., Study Chair — Universidade do Porto
Locations (2):
- Indonesian Dental Association Jl. Utan Kayu Raya no. 46 13120, Jakarta, Timur, Indonesia
- Department of Restorative Dentistry Lagos University Teaching Hospital (LUTH) Idi Araba Surulere 101014, Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: No
Results will only be presented as grouped data never as individual data.

REFERENCES:
- [Background] Kell K, Aymerich MA, Horn V. FDI-Unilever Brush Day & Night partnership: 12 years of improving behaviour for better oral health. Int Dent J. 2018 May;68 Suppl 1(Suppl 1):3-6. doi: 10.1111/idj.12404. Epub 2018 Mar 24. PMID 29573414
- [Background] Melo P, Fine C, Malone S, Frencken JE, Horn V. The effectiveness of the Brush Day and Night programme in improving children's toothbrushing knowledge and behaviour. Int Dent J. 2018 May;68 Suppl 1(Suppl 1):7-16. doi: 10.1111/idj.12410. Epub 2018 Apr 16. PMID 29660791
- [Background] Melo P, Fine C, Malone S, Horn V. Brush Day & Night Phase III to Phase IV: ensuring that good oral health habits are sustainable. Int Dent J. 2018 May;68 Suppl 1(Suppl 1):17-19. doi: 10.1111/idj.12403. Epub 2018 Mar 22. PMID 29569263
- [Background] GREENE JC, VERMILLION JR. THE SIMPLIFIED ORAL HYGIENE INDEX. J Am Dent Assoc. 1964 Jan;68:7-13. doi: 10.14219/jada.archive.1964.0034. No abstract available. PMID 14076341
- [Derived] Melo P, Malone S, Rao A, Fine C. A 21-Day School-Based Toothbrushing Intervention in Children Aged 6 to 9 Years in Indonesia and Nigeria: Protocol for a Two-Arm Superiority Randomized Controlled Trial. JMIR Res Protoc. 2020 Feb 21;9(2):e14156. doi: 10.2196/14156. PMID 32130186